CLINICAL TRIAL: NCT07037758
Title: A Phase 1b Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Tarlatamab in Combination With AB248 in Participants With Extensive Stage Small Cell Lung Cancer (DeLLphi-311)
Brief Title: A Study of Tarlatamab in Combination With AB248 in Participants With Extensive Stage Small Cell Lung Cancer (DeLLphi-311)
Acronym: DeLLphi-311
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Asher Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20240200
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Extensive Stage Small Cell Lung Cancer
Keywords: ES-SCLC; Tarlatamab; AMG 757; AB248; Imdelltra
MeSH Terms: interventions — AMG 757

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Exploration (Experimental): Multiple dose levels of AB248 will be explored in combination with tarlatamab administered via intravenous (IV) infusion.
  Interventions: Drug: Tarlatamab; Drug: AB248
- Dose Expansion (Experimental): The dose expansion part will test tarlatamab in combination with the MTCD/recommended dose for expansion of AB248 identified in the dose exploration part.
  An optional cohort may be opened based on emerging data to study tarlatamab in combination with AB248 at a lower dose than the MTCD/recommended dose for expansion or with an alternative dose regimen at a AB248 dose lower than or equal to MTCD/recommended dose for expansion.
  Interventions: Drug: Tarlatamab; Drug: AB248

INTERVENTIONS:
Drug: Tarlatamab — Administered as an IV infusion.
  Other Names: AMG 757; Imdelltra
Drug: AB248 — Administered either as an IV infusion followed by a flush or using a syringe pump without a flush.

SUMMARY:
The primary objective for dose exploration and dose expansion is to evaluate the safety and tolerability of tarlatamab in combination with AB248.

The primary objective for dose exploration only is to determine the recommended dose for expansion and/or maximum tolerated combination dose (MTCD) of AB248 in combination with tarlatamab.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided informed consent before initiation of any study-specific activities/procedures.
2. Participants ≥ 18 years (or ≥ legal age within the country if it is older than 18 years) at the time of signing the informed consent.
3. Participants with histologically or cytologically confirmed ES-SCLC that has progressed or recurred following at least 1 line of anti-cancer therapy for ES-SCLC.
4. Participants must have at least 1 measurable lesion as defined by RECIST 1.1 within 21-day screening period, not previously irradiated.
5. Participants must have adequate organ function (hematological, coagulation, cardiac, pulmonary, kidney, and liver).
6. Participants must submit a fresh tumor biopsy at screening unless a new biopsy cannot be performed safely or is infeasible. Participants who cannot provide fresh tissue may provide archival tissue that was collected after last anticancer therapy.

Exclusion Criteria:

1. Symptomatic central nervous system (CNS) metastases.
2. Participants with brain metastases may be eligible if criteria defined in the protocol are met.
3. Prior therapy with any delta-like ligand 3 (DLL3)-directed therapy (including tarlatamab).
4. Prior interleukin (IL)-2, IL-7 or IL-15 targeted therapy.
5. Baseline (at rest) requirement of supplemental oxygen.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2028-03-18 (Estimated); Study Completion 2031-01-18 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to 2.5 years
  Clinically significant changes in vital signs and clinical laboratory tests will be reported as adverse events.
Dose Exploration: Number of Participants with Dose-limiting Toxicities (DLTs) | Up to 35 days

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of Tarlatamab | Up to approximately 21 weeks
Minimum Serum Concentration (Cmin) of Tarlatamab | Up to approximately 21 weeks
Area Under the Concentration-time Curve (AUC) of Tarlatamab | Up to approximately 21 weeks
Half-life (t1/2) of Tarlatamab | Up to approximately 21 weeks
Objective Response (OR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Up to 2.5 years
Duration of Response (DOR) per RECIST 1.1 | Up to 2.5 years
Time to Response (TTR) per RECIST 1.1 | Up to 2.5 years
Disease Control (DC) per RECIST 1.1 | Up to 2.5 years
Progression-free Survival (PFS) per RECIST 1.1 | Up to 2.5 years
Time to Progression (TTP) per RECIST 1.1 | Up to 2.5 years
Time to Subsequent Therapy | Up to 2.5 years
Overall Survival (OS) | Up to 2.5 years
Number of Participants with Anti-AB248 Antibody Formation | Up to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (16):
- United States (11):
  - University of Southern California, Norris Comprehensive Cancer Center, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Norton Cancer Institute - Downtown, Louisville, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Siteman Cancer Center, St Louis, Missouri
  - Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Baptist Cancer Center, Memphis, Tennessee
  - Swedish Cancer Institute Medical Oncology, Seattle, Washington
- South Korea (2):
  - Chungbuk National University Hospital, Cheongju Chungbuk
  - Severance Hospital Yonsei University Health System, Seoul
- Turkey (Türkiye) (3):
  - Adana Sehir Egitim ve Arastirma Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com